CLINICAL TRIAL: NCT01139450
Title: Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel Group Study of 0417 Ointment
Brief Title: Study of 0417 Ointment in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0417
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — SIM0417

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Test product that contains the active pharmaceutical ingredient
  Interventions: Drug: 0417
- Reference (Active Comparator): Reference product that contains the active pharmaceutical ingredient
  Interventions: Drug: Tacrolimus Ointment 0.03%
- Vehicle (Placebo Comparator): Placebo that contains no active pharmaceutical ingredient
  Interventions: Drug: Vehicle of 0417 test product

INTERVENTIONS:
Drug: 0417 — Topical 0417 test product applied twice daily for 4 weeks
  Arms: Test
Drug: Vehicle of 0417 test product — Vehicle of 0417 test product applied twice daily for 4 weeks
  Arms: Vehicle
Drug: Tacrolimus Ointment 0.03% — Reference product for 0417 test product. Apply twice daily for 4 weeks
  Arms: Reference

SUMMARY:
The aim of this trial is to assess the efficacy of 0417 Ointment in the Treatment of Atopic Dermatitis.

Treatment medication will be administered as follows: Apply a thin layer of ointment to affected skin areas twice daily and rub in gently and completely. Study medication will be applied twice a day, approximately 12 hours apart, for approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atopic Dermatitis
* Good health with the exception of Atopic Dermatitis
* Percent Body Surface Area minimum requirements

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
* Subjects who have any systemic or dermatological disorders with the exception of Atopic Dermatitis

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fougera Pharmaceuticals Inc., Melville, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test: Test product that contains the active pharmaceutical ingredient
  Tacrolimus Ointment 0.03% test product applied twice daily for 4 weeks
- Reference: Reference product that contains the active pharmaceutical ingredient
  Protopic Ointment 0.03%, Reference product applied twice daily for 4 weeks
- Vehicle: Placebo that contains no active pharmaceutical ingredient
  Vehicle of Tacrolimus Ointment 0.03% applied twice daily for 4 weeks
Period: Overall Study
Arm/Group | Test | Reference | Vehicle
Started | 302 | 297 | 300
Completed | 275 | 272 | 262
Not Completed | 27 | 25 | 38
Not completed — Withdrawal by Subject | 7 | 10 | 13
Not completed — Lack of Efficacy | 3 | 1 | 8
Not completed — Protocol Violation | 6 | 5 | 2
Not completed — Lost to Follow-up | 9 | 7 | 11
Not completed — Administrative | 0 | 0 | 1
Not completed — Adverse Event | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Vehicle | Total
Number analyzed (Participants) | 302 | 297 | 300 | 899
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, Years | 27.74 (18.11) | 28.8 (18.99) | 27.6 (17.34) | 28.0 (18.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 194 | 186 | 566
  Male | 116 | 103 | 114 | 333
Region of Enrollment [Number; unit: participants]
  United States | 280 | 275 | 279 | 834
  Central America | 22 | 22 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Success Based on the Investigator's Global Evaluation at the End of Treatment
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Test | Reference | Vehicle
Number analyzed (Participants) | 226 | 238 | 228
participants | 123 | 130 | 86

2. Secondary Outcome: The Mean Change From Baseline in the Total Individual Clinical Signs and Symptoms Per Body Region
Time Frame: Baseline, 4 weeks

3. Secondary Outcome: The Mean Change From Baseline in Pruritus
Time Frame: Baseline, 4 weeks

4. Secondary Outcome: The Mean Change From Baseline in the Percentage Total Body Surface Affected (%BSA)
Time Frame: Baseline, 4 weeks

ADVERSE EVENTS:
Arm/Group | Test | Reference | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/302 | 0/297 | 1/300
Other Adverse Events (participants affected / at risk) | 17/302 | 12/297 | 20/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=302) | Reference (N=297) | Vehicle (N=300)
Moderate Influenza (Infections and infestations) | 1 | 0 | 0
Severe Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=302) | Reference (N=297) | Vehicle (N=300)
Application site irritation (General disorders) | 12 | 11 | 8
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 | 1 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other